CLINICAL TRIAL: NCT00593255
Title: A Multi-centre, Randomised, Parallel, Open Labelled Study to Compare the Efficiency and Safety Profile of Insulin Aspart (NovoRapid®) and Human Soluble Insulin (Novolin® R) as Meal Related Insulin in a Three Times Daily Regimen With One Injection of Novolin® N at Bedtime in Chinese Type 1 and 2 Diabetics
Brief Title: Efficacy and Safety of Insulin Aspart in Subjects With Type 1 or Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1634
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: soluble human insulin
Drug: insulin aspart
Drug: insulin NPH

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare the efficacy of postprandial plasma glucose of two treatment regimens in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes for at least 4 weeks
* Treatment with oral antidiabetic drugs (OADs) and/or insulin for at least 4 weeks
* HbA1c: 7.5-13.5%
* Body Mass Index (BMI): 18-35 kg/m2

Exclusion Criteria:

* Treatment with either soluble human insulin or insulin NPH three times daily within 3 months before trial participation
* History of drug abuse or alcohol dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2004-07; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
2-hours postprandial plasma glucose (PPPG) | after 12 weeks of treatment

SECONDARY OUTCOMES:
Percentage of subjects achieving 2-hours PPPG treatment target
Percentage of subjects achieving HbA1c treatment target
HbA1c
Fasting plasma glucose
Hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- China (3):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Harbin, Heilongjiang
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality

REFERENCES:
- [Result] Gao Y, Pan C, Zou D, Xu Z, Liu X, Guo X. Superior prandial glucose control with Insulin Aspart compared to Regular Human Insulin in Basal Bolus Therapy with NPH in Patients with Inadequately Controlled T1DM or T2DM. ADA 2006 2006; 55 (Suppl. 1): A464 (2005-PO)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com